CLINICAL TRIAL: NCT04922918
Title: Administration of Ligilactobacillus Salivarius MP101 in an Elderly Nursing Home During the COVID Pandemics
Brief Title: Ligilactobacillus Salivarius MP101 for Elderly in a Nursing Home
Acronym: PROBELDERLY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Juan M. Rodríguez, Head, Universidad Complutense de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CEIC 20/263-E_COVID
Record Dates: First submitted 2021-06-09; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: covid-19; elderly; nursing home; probiotics
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic arm (Experimental): Administration of Ligilactobacillus salivarius MP101 (>9 log10cfu, daily) for 4 months
  Interventions: Biological: Ligilactobacillus salivarius MP101

INTERVENTIONS:
Biological: Ligilactobacillus salivarius MP101 — Administration of the strain through a fermented milk

SUMMARY:
The objective of this work was to investigate the effect of Ligilactobacillus salivarius MP101 on the functional (Barthel index), cognitive (GDS/FAST) and nutritional (MNA) status, and on the nasal and fecal inflammatory profiles of elderly living in a nursing home highly affected by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Living in the nursing home
* Informed consent obtained

Exclusion Criteria:

* Absence of informed consent
* Parenteral nutrition (exclusively)
* Allergy to cow's milk protein

Ages: 74 Years to 98 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-24 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Barthel index | 4 months
  functional status score (daily activities)
MNA score | 4 months
  Nutritional status
nasal and fecal immune profile | 4 months
  37-plex

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Para Mayores Santa Isabel, S.L., Moralzarzal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No